CLINICAL TRIAL: NCT06836596
Title: Efficacy of Sensory Electrical Stimulation Versus Alternating Electromyogram (EMG) On Functional Recovery Of Hand in Chronic Stroke Survivors :Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez University (Other)
Responsible Party: Principal Investigator, Dany Alphonse Anwar Habib, Lecturer of Physical Therapy for Neurology and Its Surgery, Suez University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/004916
Record Dates: First submitted 2025-02-15; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Chronic Stroke Survivors; Chronic Stroke Survivors With Plegic Hand
Keywords: Sensory Electrical Stimulation - Alternating Electromyogram (EMG) - Functional Recovery - Hand - Chronic Stroke Survivors
MeSH Terms: interventions — Electromyography

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Sensory Electrical Stimulation Group) (Experimental): This group receives the active treatment of peripheral sensory electrical stimulation along with the hand function training program, making it the experimental group being tested for its effects on improving hand function in stroke patients.
  Interventions: Device: Peripheral sensory electrical stimulation via Elettronica Pagani Roland series model: ET 20 S/N: 1907 (Made in Italy)
- Group B (Alternating EMG Stimulation Group) (Active Comparator): This is because this group is receiving a different active treatment (alternating EMG stimulation) along with hand function training, and it is being compared to the other active treatment (sensory electrical stimulation) in Group A. Both groups are experimental, but Group B serves as a comparison to Group A in the study.
  Interventions: Device: Alternating electromyogram (EMG) neuromuscular electrical stimulation via MyoTrac Infiniti device (T9800, Thought Technology Ltd. Montreal, Quebec, Canada)
- Group C (Control Group) (No Intervention): Group C only receives the designed hand function training program and does not receive any form of electrical stimulation, the electrodes are used, but no active stimulation is delivered. It serves as the control group for comparison against the experimental treatments in Groups A and B.

INTERVENTIONS:
Device: Peripheral sensory electrical stimulation via Elettronica Pagani Roland series model: ET 20 S/N: 1907 (Made in Italy) — Sensory electrical stimulation, Transcutaneous electrical nerve stimulation (TENS) involves delivering electrical current through electrodes placed on the skin to manage pain. It can be applied at different frequencies, ranging from low (50 Hz). The intensity can be adjusted from sensory to motor levels. Sensory intensity is when the patient experiences a strong yet comfortable sensation without triggering muscle contraction
  Arms: Group A (Sensory Electrical Stimulation Group)
Device: Alternating electromyogram (EMG) neuromuscular electrical stimulation via MyoTrac Infiniti device (T9800, Thought Technology Ltd. Montreal, Quebec, Canada) — the device detects the EMG threshold value (peak muscle torque) of the target muscle and activates stimulation to enhance the patient's voluntary activation of the targeted muscle groups. It is used to assess peak muscle torque and deliver alternating and EMG-triggered stimulation. Surface electrodes are employed to detect electromyography in the affected muscle and administer electrical stimulation to the targeted muscle during treatment. The device stimulates the targeted muscles, after which the patient attempts to replicate the same movement until reaching the preset EMG feedback level
  Arms: Group B (Alternating EMG Stimulation Group)

SUMMARY:
This study aims to find out which treatment works better for improving hand function in stroke patients: sensory electrical stimulation or alternating electromyogram (EMG) stimulation. Both methods use electrical stimulation to help patients regain hand movement, but they work in slightly different ways. The goal is to see if one method is more effective than the other in helping stroke survivors recover their hand abilities.

ELIGIBILITY:
Inclusion Criteria:

* Chronic stroke patients were between 45 and 65 years old, with a duration of illness ranging from 6 to 18 months post-stroke. They exhibited upper extremity spasticity no greater than 1+ on the Modified Ashworth Scale. Patients were cooperative, as indicated by a Mini-Mental State Examination (MMSE) score of ≥ 24, and were capable of grasping and releasing at least one block in the Box and Block Test.

Exclusion Criteria:

* Hand function impairment caused by factors other than stroke, unstable health conditions such as cardiac dysfunction, end-stage renal failure, or uncontrolled diabetes, long-term use of medications that may affect motor or sensory excitability, contractures or restrictions in wrist joint range of motion, pre-existing musculoskeletal diseases significantly impacting physical function, and a history of Botulinum Toxin injection in the hand muscles.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-12-07 (Actual); Study Completion 2025-02-07 (Actual)

PRIMARY OUTCOMES:
Action Research Arm Test (ARAT) | 12 weeks
  assessment tool to evaluate the hand and arm function in individuals with stroke. It is often used to measure improvements in motor function, particularly for tasks like grasping, gripping, and other fine motor skills. It consists of 19 items assessing different aspects of arm and hand function, including tasks like reaching, grasping, and lifting objects. These tasks are scored, and the total score reflects the level of motor recovery and functional ability.
modified Ashworth scale | 12 weeks
  is a widely used tool to assess spasticity, or increased muscle tone, in individuals with neurological conditions like stroke. It measures the resistance of a muscle to passive movement and helps evaluate the degree of spasticity in the affected limbs. MAS Scoring (for elbow, wrist, and shoulder): 0: No increase in muscle tone. 1: Slight increase in muscle tone, manifested by a catch and release or minimal resistance at the end of the range of motion.
  1+: Slight increase in muscle tone, manifested by a catch followed by minimal resistance throughout the remainder of the range of motion.
  2: More marked increase in muscle tone through most of the range of motion, but the affected part(s) can still be easily moved.
  3: Considerable increase in muscle tone, making passive movement difficult. 4: Affected part(s) rigid in flexion or extension.
Medical Research Council scale for Fingers and Wrist | 12 weeks
  The Medical Research Council (MRC) Scale is a widely used method to assess muscle strength in different muscle groups, and to evaluate the strength of the fingers and wrist in stroke patients as part of this study.
  The MRC Scale is a 6-point grading system used to measure muscle strength. Grade 0: No contraction - There is no visible or palpable muscle contraction. Grade 1: Trace contraction - A slight contraction can be felt, but no movement occurs.
  Grade 2: Active movement, but not against gravity - The muscle can move the joint, but not against gravity.
  Grade 3: Active movement against gravity - The muscle can move the joint against gravity but not against resistance.
  Grade 4: Active movement against some resistance - The muscle can move the joint against resistance but is weaker than normal strength.
  Grade 5: Normal strength - The muscle can move the joint against full resistance with no weakness.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy, Cairo universuty, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No
because they are Potential for Misuse. I am concerned about the misuse of IPD, where the data could be used to advance conflicting interests, such as in studies that are biased toward certain results or that could be manipulated to serve commercial purposes